CLINICAL TRIAL: NCT03848494
Title: True Short Esophagus in Gastroesophageal Reflux Disease or Hiatus Hernia
Brief Title: True Short Esophagus in Gastroesophageal Reflux Disease
Status: Completed | Type: Observational
Sponsor: University of Bologna (Other)
Responsible Party: Principal Investigator, Marialuisa Lugaresi, Adjunct Professor MD, PhD, University of Bologna
Other Study IDs: True Short Esophagus-2019
Record Dates: First submitted 2019-01-23; First posted 2019-02-20 (Actual); Last update posted 2019-02-20 (Actual); Status verified 2019-02

CONDITIONS: Gastroesophageal Reflux Disease
Keywords: gastroesophageal reflux disease; hiatus hernia
MeSH Terms: conditions — Gastroesophageal Reflux; Hernia, Hiatal | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Gastroesophageal reflux disease: Patients submitted to primary minimally invasive surgery for gastroesophageal reflux disease or hiatus hernia
  Interventions: Procedure: Surgery

INTERVENTIONS:
Procedure: Surgery — Laparoscopic floppy Nissen, laparoscopic-left thoracoscopic Collis-Nissen, laparoscopic gastric fundus wrapped around the stomach

SUMMARY:
True short esophagus is controversial in surgery for gastroesophageal reflux disease and hiatus hernia. Recently, it was published that extensive esophageal mobilization achieved an esophageal length adequate to perform around the esophagus fundoplication in all cases with satisfactory long-term results.

DETAILED DESCRIPTION:
In the 1960s, surgery for hiatus hernia and gastroesophageal reflux disease were introduced based on anatomical principles. The technical foundations of the new surgery were essentially dictated by experience. The following findings were reported: the stomach must be wrapped around an adequate segment of intra-abdominal esophagus, the antireflux barrier is efficient if the fundoplication acts under abdominal pressure and tension over sutures must be minimal to avoid disruption. Since the early use of open antireflux surgery, controversy has arisen between surgeons who treat patients using dedicated techniques in cases diagnosed with a shortened esophagus and surgeons who deny the existence of short esophagus. The clinical results achieved by both parties were not different, independently of the adoption of an open or minimally invasive technique. In 2008, a multicenter study found that true short esophagus was present in almost 20% of patients who were routinely submitted to surgery for gastroesophageal reflux disease and/or not axial hiatus hernias; the study was based on intraoperative measurements obtained in centimeters of the distance between the gastric folds considered the gastroesophageal junction and the apex of the diaphragm after extensive mobilization of the intra thoracic esophagus. Recently, in a study performed to assess symptomatic recurrence in patients who underwent laparoscopic repair of large hernias, the authors did not perform any esophageal lengthening procedures because an adequate segment of abdominal esophagus was always achieved after extended esophageal mobilization; they concluded that the use of proton pump inhibitors for the medical management of gastroesophageal reflux disease may have reduced the formation of peptic stricture, which is associated with short esophagus, and that esophageal lengthening procedures should probably no longer be applied.

In this study, the position of the gastroesophageal junction with respect for the diaphragmatic hiatus was assessed subjectively. Once more, crucial questions related to the debate on short esophagus were raised: is it possible that a) without an objective assessment of the position of the gastroesophageal junction , the gastric fundus may be inadvertently wrapped around the hypo cardia stomach, which acquires a tubular shape as a consequence of progressive esophageal shortening; and b) can the unconventional stomach around stomach fundoplication approach achieve good clinical results? To answer these questions, the investigators considered cases operated upon to gastroesophageal reflux disease and hiatus hernia since 2004, when was routinely adopted the use of intraoperative endoscopic assessment of the gastroesophageal junction position with respect for the diaphragmatic hiatus, were considered. In this series, participants were grouped according to the radiological classification of hiatus hernia, the length of the intra-abdominal esophagus, the surgical techniques adopted.

ELIGIBILITY:
Inclusion Criteria:

* Patients submitted to primary minimally invasive surgery for gastroesophageal reflux diseases or hiatus hernia.
* Age > 18 years.

Exclusion Criteria:

* Patients already submitted to minimally invasive surgery for gastroesophageal reflux diseases or hiatus hernia for recurrence of the disease.
* Patients submitted to open surgery for gastroesophageal reflux diseases or hiatus hernia.
* Patients affected by other esophageal diseases.
* Age < 18 years.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients affected by gastroesophageal reflux disease or hiatus hernia submitted to primary minimally invasive surgery.
Sampling Method: Probability Sample
Enrollment: 311 (Actual)
Dates: Start 2004-01-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Frequency of true short esophagus | 9 years
  Intraoperative abdominal esophageal length < 1.5 cm
Long term results after surgery | 9 years
  Excellent = no reflux symptoms or dysphagia or esophagitis; good = slight reflux symptoms or dysphagia on a monthly basis and no esophagitis; fair = moderate reflux symptoms or dysphagia on a weekly basis; grade A esophagitis according to Los Angeles classification; poor = severe reflux symptoms or dysphagia on a daily basis and esophagitis B,C,D according to Los Angeles classification.

CONTACTS AND LOCATIONS:
Overall Officials: Marialuisa Lugaresi, MD, PhD, Principal Investigator — Department of Medical and Surgical Sciences University of Bologna Italy

IPD SHARING:
Plan to Share IPD: No